CLINICAL TRIAL: NCT05734053
Title: Nilotinib for Patients With Chronic Myeloid Leukemia in First Line and Any Subsequent Line - a Non-interventional Study on the Assessment of Deep Molecular Response in CML Patients in Daily Routine.
Brief Title: Nilotinib for Patients With Chronic Myeloid Leukemia in First Line and Any Subsequent Line
Acronym: NOFRETETE
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAMN107ADE23
Record Dates: First submitted 2023-02-09; First posted 2023-02-17 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic myeloid leukemia; CML; NOFRETETE; Nilotinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Nilotinib: patients prescribed with nilotinib in routine medical practice
  Interventions: Other: Nilotinib

INTERVENTIONS:
Other: Nilotinib — There was no treatment allocation. Patients administered Nilotinib by prescription could be enrolled.
  Other Names: Tasigna

SUMMARY:
This was a non-interventional observational study within the routine chronic myeloid leukemia treatment practice; no further tests were required apart from the assessments routinely performed for Chronic myeloid leukemia patients treated with nilotinib.

DETAILED DESCRIPTION:
The observation period per patient was 24 months. All patients were treated with nilotinib in accordance to the clinical routine at the respective institution and the summary of product characteristics (SmPC).

The observation intervals (documentation at baseline and at about 3, 6, 9, 12, 18 and 24 months) were not fixed and were aligned with the regular treatment schedule and the clinical symptoms of each patient. The medical decision about the schedule as well as therapeutic and diagnostic measures was made solely by the responsible physician. Patients who discontinued treatment within two years of the observation period were followed until starting a new TKI therapy line, however with a maximum time period of six months. All other patients that reached the official end of treatment after completion of the 24-month observation period were followed up for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with Ph+ CML (or evidence of BCR-ABL transcript) treated with nilotinib under routine medical practice and the SmPC, as amended, in first or any subsequent line, if the current therapy with nilotinib has not been in place for more than twelve months. Retrospective documentation of patients for up to one year will be permitted.
* Patients who have already had an interruption/discontinuation of nilotinib therapy.
* Patients who have been informed about this NIS and have personally dated and signed their informed consent form.

Exclusion Criteria:

* There are no exclusion criteria, apart from the contraindications mentioned in the SmPC. Participating patients are not allowed to take part in a clinical trial in parallel,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male and female patients with diagnosed Philadelphia chromosome positive (Ph+) and/or Breakpoint cluster region-Abelson tyrosine kinase (Abelson murine leukemia proto-oncogene)+ Chronic myeloid leukemia who were being treated with nilotinib in first or any subsequent line and for whom treatment with nilotinib was indicated according to SmPC
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2016-06-28 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-09-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in Major molecular response (MMR), and Deep molecular response according to international standard (MR^4.0 and MR^4.5) | 24 months
  Proportion of patients in MMR, MR^4.0 and MR^4.5 was collected
Time to achievement of an MR4.0 and MR4.5 | 24 months
  Time to achievement of an MR4.0 and MR4.5 was collected
Duration of an MR4.0 and MR4.5 | 24 months
  Duration of an MR4.0 and MR4.5 was collected
Proportion of patients whose molecular response is routinely analyzed by a MR4.5-certified laboratory | 24 months
  Proportion of patients whose molecular response is routinely analyzed by a MR4.5-certified laboratory was collected
Proportion of European Treatment and Outcome Study for CML (EUTOS)-qualified laboratories that perform qRT-PCR. | 24 months
  Proportion of European Treatment and Outcome Study for CML (EUTOS)-qualified laboratories that perform qRT-PCR was documented
Patient-reported QoL | 24 months
  The EORTC QLQ-C30 questionnaire in conjunction with the EORTC QLQ-CML24 module was used to assess patient-reported QoL.
Patient adherence | 24 months
  Patient adherence was documented using the MMAS-8 (Morisky et al., 2008) patient questionnaire.
Proportion of patients who discontinue Tyrosine kinase inhibitor (TKI) therapy | 24 months
  Proportion of patients who discontinue Tyrosine kinase inhibitor (TKI) therapy was documented

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (71):
- Germany (71):
  - Novartis Investigative Site, Freudenstadt, Baden-Wurttemberg
  - Novartis Investigative Site, Aschaffenburg, Bavaria
  - Novartis Investigative Site, Augsburg, Bavaria
  - Novartis Investigative Site, Bayreuth, Bavaria
  - Novartis Investigative Site, Coburg, Bavaria
  - Novartis Investigative Site, Donauwörth, Bavaria
  - Novartis Investigative Site, Kronach, Bavaria
  - Novartis Investigative Site, Landshut, Bavaria
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Frankfurt (Oder), Brandenburg
  - Novartis Investigative Site, Baden-Württemberg, Heidenheim a.d.B
  - Novartis Investigative Site, Erbach im Odenwald, Hesse
  - Novartis Investigative Site, Goslar, Lower Saxony
  - Novartis Investigative Site, Göttingen, Lower Saxony
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Twistringen, Lower Saxony
  - Novartis Investigative Site, Westerstede, Lower Saxony
  - Novartis Investigative Site, Aachen, North Rhine-Westphalia
  - Novartis Investigative Site, Neuss, North Rhine-Westphalia
  - Novartis Investigative Site, Ahaus, Northrhine Westfalia
  - Novartis Investigative Site, Bad Salzuflen, Northrhine Westfalia
  - Novartis Investigative Site, Hagen, Northrhine Westfalia
  - Novartis Investigative Site, Iserlohn, Northrhine Westfalia
  - Novartis Investigative Site, Neuwied, Rhineland-Palatinate
  - Novartis Investigative Site, Bad Schlema, Saxony
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Zittau, Saxony
  - Novartis Investigative Site, Reinbek, Schleswig-Holstein
  - Novartis Investigative Site, Altötting
  - Novartis Investigative Site, Bad Liebenwerda
  - Novartis Investigative Site, Bad Mergentheim
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Biberach
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Halberstadt
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hamelin
  - Novartis Investigative Site, Hamm
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heilbronn
  - Novartis Investigative Site, Hildesheim
  - Novartis Investigative Site, Lemgo
  - Novartis Investigative Site, Ludwigsburg
  - Novartis Investigative Site, Memmingen
  - Novartis Investigative Site, Merseburg
  - Novartis Investigative Site, Moers
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Neumünster
  - Novartis Investigative Site, Nordhorn
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Offenburg
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Porta Westfalica
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Rotenburg (Wümme)
  - Novartis Investigative Site, Rüsselsheim am Main
  - Novartis Investigative Site, Schorndorf
  - Novartis Investigative Site, Singen
  - Novartis Investigative Site, Speyer
  - Novartis Investigative Site, Stolberg
  - Novartis Investigative Site, Viersen
  - Novartis Investigative Site, Wiesbaden
  - Novartis Investigative Site, Wilhelmshaven
  - Novartis Investigative Site, Wolfsburg
  - Novartis Investigative Site, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for Study CAMN107ADE23 that is getting linked from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18084